CLINICAL TRIAL: NCT01585779
Title: Contour 3D®/TriAd® Tricuspid Annuloplasty Ring Post-Market Clinical Trial
Acronym: Contour3D
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: 10030481DOC
Record Dates: First submitted 2012-04-18; First posted 2012-04-26 (Estimated); Results first posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Tricuspid Valve Regurgitation; Tricuspid Valve Insufficiency
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Contour 3D® Implant: The subject population includes patients indicated for a TV repair procedure concomitant to left-sided heart surgery, and for whom the surgeon considers the implantation of a Contour 3D® ring most appropriate to reconstruct the diseased valve. Patients with primary TV regurgitation will not be included in this study. Implantation with the Contour 3D® ring will occur in conjunction with another concomitant surgical repair procedure
  Interventions: Device: Contour 3D® implant for tricuspid valve repair
- Tri-Ad® Implant: The subject population includes patients indicated for a TV repair procedure concomitant to left-sided heart surgery, and for whom the surgeon considers the implantation of a Tri-Ad® ring most appropriate to reconstruct the diseased valve. Patients with primary TV regurgitation will not be included in this study. Implantation with the Tri-Ad® ring will occur in conjunction with another concomitant surgical repair procedure
  Interventions: Device: Tri-Ad® implant for tricuspid valve repair

INTERVENTIONS:
Device: Contour 3D® implant for tricuspid valve repair — Tricuspid annuloplasty ring
  Groups: Contour 3D® Implant
Device: Tri-Ad® implant for tricuspid valve repair — Tricuspid annuloplasty ring
  Groups: Tri-Ad® Implant

SUMMARY:
The purpose of this study is to gather clinical information on the hemodynamic performance of the Contour 3D® and Tri-Ad® Tricuspid Annuloplasty Rings in a post-market environment.

DETAILED DESCRIPTION:
The primary goal of the TV repair procedure is to relieve patients from TV insufficiency or reduce TV stenosis. This study will evaluate the hemodynamic efficacy of the Contour 3D® and Tri-Ad® ring and characterize the effect of the TV repair through assessment of right atrial size and right ventricular function. Additionally, this study will characterize the patient population for whom a Contour 3D® or Tri-Ad® ring is chosen to repair TV insufficiency. Health status and adverse events (AE) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Subject or legal guardian willing and able to sign and date the Informed Consent Form (and Authorization to Use and Disclose Health Information Form, if applicable)
* Subject indicated for a concomitant surgical repair of the TV
* Subject is willing to return for required follow-up visits to the hospital where the implantation originally occurred

Exclusion Criteria:

* Subject with a degenerative TV condition
* Subject with primary TV regurgitation
* Subject with a previous TV repair or replacement
* Subject indicated for a stand-alone TV repair
* Subject currently participating in an investigational drug or another device study
* Subject with life expectancy of less than one year
* Subject is pregnant or desires to be pregnant within 12 months following implantation
* Subject is under 18 or over 85 years of age
* Subject with active endocarditis
* Subject with valvular retraction with severely reduced mobility
* Subject with a heavily calcified TV

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population includes patients indicated for a TV repair procedure concomitant to left-sided heart surgery, and for whom the surgeon considers the implantation of a Contour 3D® or Tri-Ad® ring most appropriate to reconstruct the diseased valve. Patients with primary TV regurgitation will not be included in this study. Implantation with the Contour 3D® or Tri-Ad® ring will occur in conjunction with another concomitant surgical repair procedure
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2012-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Vang, Study Director — Medtronic
Locations (3):
- United States (3):
  - Florida Heart & Vascular Care at Aventura, Aventura, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Mission Hospital Research Institute, Asheville, North Carolina

REFERENCES:
- See also: Sponsor website — http://www.medtronic.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Started | 36 | 28
Completed | 26 | 21
Not Completed | 10 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant | Total
Number analyzed (Participants) | 36 | 28 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 3 | 16
  >=65 years | 23 | 25 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (11.6) | 73.7 (8.5) | 70.7 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 33
  Male | 21 | 10 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in the Degree of Tricuspid Regurgitation
Description: The primary objective is the evaluation of hemodynamic performance of the TV postimplant of a tricuspid annuloplasty ring in a postmarket environment.
  Degree of TV regurgitation - Change in the degree of tricuspid regurgitation from preimplant through 12 months postimplant.
Time Frame: Preimplant through Discharge
Measure: Number; unit: participants
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Number analyzed (Participants) | 35 | 25
participants
  Improved | 27 | 18
  No Change | 6 | 6
  Worsened | 2 | 1

2. Primary Outcome: Change in the Degree of Tricuspid Regurgitation
Description: as for outcome 1
Time Frame: Preimplant through 6 Months
Measure: Number; unit: participants
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Number analyzed (Participants) | 30 | 20
participants
  Improved | 23 | 14
  No Change | 6 | 4
  Worsened | 1 | 2

3. Primary Outcome: Change in the Degree of Tricuspid Regurgitation
Description: as for outcome 1
Time Frame: Preimplant through 12 Months
Measure: Number; unit: participants
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Number analyzed (Participants) | 25 | 20
participants
  Improved | 17 | 12
  No Change | 5 | 7
  Worsened | 3 | 1

4. Primary Outcome: The Mean Gradient Across the Tricuspid Valve
Description: The primary objective is the evaluation of hemodynamic performance of the TV postimplant of a tricuspid annuloplasty ring in a postmarket environment by analysis of the mean gradient across the tricuspid valve. The mean gradient across the tricuspid valve measured at discharge, 6 months, and 12 months post-implant
Time Frame: Discharge
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Number analyzed (Participants) | 35 | 26
mmHg | 2.2 [1.9 to 3.0] | 2.0 [2.0 to 3.0]

5. Primary Outcome: The Mean Gradient Across the Tricuspid Valve
Description: as for outcome 4
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Number analyzed (Participants) | 30 | 20
mmHg | 2.0 [1.3 to 3.0] | 2.2 [1.6 to 3.0]

6. Primary Outcome: The Mean Gradient Across the Tricuspid Valve
Description: as for outcome 4
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Number analyzed (Participants) | 25 | 21
mmHg | 2.0 [1.9 to 3.0] | 2.0 [1.0 to 2.0]

7. Primary Outcome: Change in the Degree of TV Leaflet Coaptation Length
Description: The primary objective is the evaluation of hemodynamic performance of the TV postimplant of a tricuspid annuloplasty ring in a postmarket environment by analysis of the TV leaflet coaptation length. Change in the degree of TV leaflet coaptation length from preimplant through 12 months postimplant.
Time Frame: Preimplant through Discharge
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Number analyzed (Participants) | 34 | 24
mm | 0.0 [-2.9 to 2.0] | 0.0 [-1.0 to 1.8]

8. Primary Outcome: Change in the Degree of TV Leaflet Coaptation Length
Description: as for outcome 7
Time Frame: Preimplant through 6 Months
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Number analyzed (Participants) | 29 | 19
mm | 1.0 [-1.0 to 2.0] | 0.0 [-2.1 to 1.0]

9. Primary Outcome: Change in the Degree of TV Leaflet Coaptation Length
Description: as for outcome 7
Time Frame: Preimplant through 12 Months
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Number analyzed (Participants) | 25 | 20
mm | 0.0 [-2.0 to 1.0] | 0.0 [-2.1 to 1.0]

10. Primary Outcome: Change in the Degree of TV Leaflet Tethering Height
Description: The primary objective is the evaluation of hemodynamic performance of the TV postimplant of a tricuspid annuloplasty ring in a postmarket environment by analysis of the TV leaflet tethering height. Change in the degree of TV leaflet tethering height from pre-implant through 12 months post-implant.
Time Frame: Preimplant through Discharge
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Number analyzed (Participants) | 34 | 24
mm | -0.8 [-2.0 to 1.0] | 0.5 [-0.6 to 2.0]

11. Primary Outcome: Change in the Degree of TV Leaflet Tethering Height
Description: as for outcome 10
Time Frame: Preimplant through 6 Months
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Number analyzed (Participants) | 29 | 19
mm | 0.6 [-2.0 to 3.0] | 1.0 [-1.0 to 2.0]

12. Primary Outcome: Change in the Degree of TV Leaflet Tethering Height
Description: as for outcome 10
Time Frame: Preimplant through 12 Months
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Number analyzed (Participants) | 25 | 20
mm | 1.0 [-1.0 to 2.5] | 1.0 [-2.7 to 3.0]

13. Secondary Outcome: Change in the Right Ventricle (RV) Diastolic Area
Description: The secondary objective is the evaluation of effect of TV repair with the study ring on Right ventricle (RV) diastolic area at end diastole. Change in the Right ventricle (RV) diastolic area from preimplant through 12 months post-implant.
Time Frame: Preimplant through Discharge
Measure: Median (Inter-Quartile Range); unit: mm^2
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Number analyzed (Participants) | 31 | 22
mm^2 | -140.0 [-585.0 to 61.0] | 141.0 [-492.0 to 561.0]

14. Secondary Outcome: Change in the Right Ventricle (RV) Diastolic Area
Description: as for outcome 13
Time Frame: Preimplant through 6 Months
Measure: Median (Inter-Quartile Range); unit: mm^2
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Number analyzed (Participants) | 28 | 17
mm^2 | 160.5 [-155.0 to 451.0] | 70.6 [-374.0 to 499.0]

15. Secondary Outcome: Change in the Right Ventricle (RV) Diastolic Area
Description: as for outcome 13
Time Frame: Preimplant through 12 Months
Measure: Median (Inter-Quartile Range); unit: mm^2
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Number analyzed (Participants) | 24 | 18
mm^2 | 395.0 [-12.5 to 626.5] | 211.0 [-174.0 to 550.0]

16. Secondary Outcome: Change in the Tricuspid Annular (Basal) Diameter
Description: The secondary objective is the evaluation of effect of TV repair with the study ring on Tricuspid annular (basal) diameter. Change in the tricuspid annular (basal) diameter from preimplant through 12 months post-implant
Time Frame: Preimplant through Discharge
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Number analyzed (Participants) | 34 | 23
mm | -4.0 [-6.0 to 2.0] | 0.0 [-4.0 to 6.0]

17. Secondary Outcome: Change in the Tricuspid Annular (Basal) Diameter
Description: as for outcome 16
Time Frame: Preimplant through 6 Months
Measure: Median (Inter-Quartile Range); unit: mm
Groups:
- Tri-Ad® Implant: The subject population includes patients indicated for a TV repair procedure concomitant to left-sided heart surgery, and for whom the surgeon considers the implantation of a Tri-Ad® ring most appropriate to reconstruct the diseased valve. Patients with primary TV regurgitation will not be included in this study. Implantation with the Tri-Ad® ring will occur in conjunction with another concomitant surgical repair procedure Tri-Ad® implant for tricuspid valve repair: Tricuspid annuloplasty ring
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Number analyzed (Participants) | 29 | 18
mm | 3.0 [-4.0 to 7.0] | 1.0 [-8.0 to 6.0]

18. Secondary Outcome: Change in the Tricuspid Annular (Basal) Diameter
Description: as for outcome 16
Time Frame: Preimplant through 12 Months
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Number analyzed (Participants) | 25 | 19
mm | 4.0 [-2.0 to 7.0] | 1.0 [-6.0 to 11.0]

19. Secondary Outcome: Change in the RV Fractional Area
Description: The secondary objective is the evaluation of effect of TV repair with the study ring on RV fractional area. Change in the RV fractional area preimplant through 12 months post-implant.
Time Frame: Preimplant through Discharge
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Number analyzed (Participants) | 31 | 22
percent | -3.8 [-15.6 to 4.0] | -1.8 [-14.3 to 11.8]

20. Secondary Outcome: Change in the RV Fractional Area
Description: as for outcome 19
Time Frame: Preimplant through 6 Months
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Number analyzed (Participants) | 28 | 17
percent | -0.8 [-10.0 to 7.2] | -6.2 [-12.9 to 3.8]

21. Secondary Outcome: Change in the RV Fractional Area
Description: as for outcome 19
Time Frame: Preimplant through 12 Months
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Number analyzed (Participants) | 24 | 18
percent | -0.4 [-12.2 to 7.9] | -3.6 [-13.4 to 0.3]

22. Secondary Outcome: Demographic Data
Description: Characterize the patient population for which an annuloplasty ring is chosen to repair TV insufficiency and assess the effect of TV repair with the study ring on the tricuspid valve functional status
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Number analyzed (Participants) | 36 | 28
participants
  Previous Valve Repair | 5 | 1
  Previous Valve Replacement | 2 | 3
  Previous CABG | 6 | 5
  CAD | 12 | 15
  CHF | 19 | 13
  Atrial Fibrillation/flutter | 22 | 18
  MI | 4 | 4
  Diabetes | 11 | 6
  Hypertension | 27 | 24
  Moderate or severe aortic valve insufficiency | 3 | 3
  Moderate or severe mitral valve insufficiency | 31 | 23

23. Secondary Outcome: Change in New York Heart Association (NYHA) Classification
Description: Assess the effect of TV repair with the study ring on the tricuspid valve functional status by analysis of the New York Heart Association (NYHA) classification from pre-implant through 12 months post-implant.
Time Frame: Preimplant through Discharge
Measure: Number; unit: participants
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Number analyzed (Participants) | 36 | 26
participants
  Improved | 19 | 15
  No Change | 13 | 6
  Worsened | 4 | 5

24. Secondary Outcome: Change in New York Heart Association (NYHA) Classification
Description: as for outcome 23
Time Frame: Preimplant through 6 months
Measure: Number; unit: participants
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Number analyzed (Participants) | 30 | 21
participants
  Improved | 20 | 19
  No Change | 8 | 1
  Worsened | 2 | 1

25. Secondary Outcome: Change in New York Heart Association (NYHA) Classification .
Description: as for outcome 23
Time Frame: Preimplant through 12 months
Measure: Number; unit: participants
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Number analyzed (Participants) | 26 | 21
participants
  Improved | 19 | 17
  No Change | 7 | 3
  Worsened | 0 | 1

ADVERSE EVENTS:
Time Frame: Device or procedure related Adverse events (AEs) were collected from study enrollment to study closure, up to 1 year.
Description: All new or worsening device or procedure related AEs were collected through1 year.
Arm/Group | Contour 3D® Implant | Tri-Ad® Implant
Serious Adverse Events (participants affected / at risk) | 16/36 | 10/28
Other Adverse Events (participants affected / at risk) | 2/36 | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Contour 3D® Implant (N=36) | Tri-Ad® Implant (N=28)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (3) | 3 (3)
Atrioventricular block complete (Cardiac disorders) | 2 (2) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery embolism (Cardiac disorders) | 1 (1) | 0 (0)
Nodal rhythm (Cardiac disorders) | 1 (1) | 2 (2)
Sinus node dysfunction (Cardiac disorders) | 2 (2) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac output decreased (Investigations) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (2)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 3 (3) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Contour 3D® Implant (N=36) | Tri-Ad® Implant (N=28)
Atrioventricular block first degree (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days